CLINICAL TRIAL: NCT03385265
Title: An Interactive mHealth App for Better Glycemic Control in Parents of Young Kids With T1D
Brief Title: Iterative Beta Testing of Videos for the DIPPer Academy
Acronym: DIPPer Academy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15040153; 1DP3DK108211-01 (NIH)
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIPPer Academy (Experimental): Parents randomized to this group will participate in the DIPPer Academy curriculum.
  Interventions: Behavioral: DIPPer Academy
- Standard of Care Control (Active Comparator): Parents randomized to this group will receive care as usual from their child's diabetes provider
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: DIPPer Academy — The DIPPer Academy curricula will build on treatment models guided by the Health Beliefs Model (HBM) and Social Cognitive Theory (SCT). The curricula includes video microlectures, personalize progress reports, and other features delivered via the internet.
  Arms: DIPPer Academy
Other: Standard of Care — Parents in the standard of care control group will be instructed to manage their child's T1D as recommended by the diabetes team.
  Arms: Standard of Care Control

SUMMARY:
The purpose of this research is to develop DIPPer Academy, a parent-focused, mobile health (mHealth) behavioral intervention to promote glycemic control in young children.

DETAILED DESCRIPTION:
Because many young children with T1D have glucose levels that exceed targets, investigators need to develop efficacious, accessible, and readily disseminable interventions to help them to improve their glycemic control. To do this, the investigators need efficacious interventions that specifically address the challenges that parents of young children face in daily T1D management. Providers need mHealth interventions that minimize barriers that parents experience when trying to access face-to-face or in clinic interventions. Finally, interventions are needed that are packaged to be easily deployable by other diabetes centers. The investigator's proposed intervention, DIPPer Academy, will include all of these recommended advancements.

ELIGIBILITY:
Inclusion Criteria:

* Parents of a young child who is between 3-5.99 years old and at least 6 months post T1D diagnosis
* Parents who are English-speaking.

Exclusion Criteria:

* Parents of young children with evidence of type 2 diabetes or monogenic diabetes.
* Parents with evidence of severe psychiatric disorder.
* Parents of young children with a comorbid chronic illness (e.g., renal disease) that requires ongoing care beyond T1D.
* Parents of young children with a history of anemia or medication use that may interact with glycemic control (e.g., systemic steroids).

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve-Lynn Nelson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Children's Mercy Hospital, Kansas City, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited in clinic or by telephone.
Pre-assignment Details: pre-assignment all parents completed baseline assessment measures
Groups:
- DIPPer Academy- Parents: Parents randomized to this group will participate in the DIPPer Academy curriculum via the internet.
- Standard of Care Control- Parents: Standard of Care: Parents in the standard of care control group will be instructed to manage their child's T1D as recommended by their diabetes team.
- DIPPer Academy- Children: Parents randomized to this group will participate in DIPPer Academy via the internet. We collect Child HbA1c levels. Children do not receive treatment.
- Standard of Care- Children: Standard of Care: Parents in the standard of care control group will be instructed to manage their child's T1D as recommended by their diabetes team. We collect Child HbA1c levels.
Period: Overall Study
Arm/Group | DIPPer Academy- Parents | Standard of Care Control- Parents | DIPPer Academy- Children | Standard of Care- Children
Started | 20 | 11 | 20 | 11
Completed | 15 (this is Time 3 or 33 weeks post-baseline) | 9 (this is Time 3 or 33 weeks post-baseline) | 15 (this is Time 3 or 33 weeks post-baseline) | 9 (this is Time 3 or 33 weeks post-baseline)
Not Completed | 5 | 2 | 5 | 2
Not completed — Withdrawal by Subject | 5 | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Population: overall baseline participant number is consistent with flow documentation
Groups:
- DIPPer Academy- Parents: Parents randomized to this group will participate in the DIPPer Academy curriculum.
  DIPPer Academy: The DIPPer Academy curricula will build on treatment models guided by the Health Beliefs Model (HBM) and Social Cognitive Theory (SCT). The curricula includes video microlectures, personalize progress reports, and other features delivered via the internet.
- DIPPer Academy- Children: Parents randomized to this group will participate in the DIPPer Academy curriculum. We collect children's HbA1c level.
  DIPPer Academy: The DIPPer Academy curricula will build on treatment models guided by the Health Beliefs Model (HBM) and Social Cognitive Theory (SCT). The curricula includes video microlectures, personalize progress reports, and other features delivered via the internet. Children do not receive treatment.
- Standard of Care Control- Children: Standard of Care: Parents in the standard of care control group will be instructed to manage their child's T1D as recommended by their diabetes team. We collect children's HbA1c level.
- Total: Total of all reporting groups
Arm/Group | DIPPer Academy- Parents | Standard of Care Control- Parents | DIPPer Academy- Children | Standard of Care Control- Children | Total
Number analyzed (Participants) | 20 | 11 | 20 | 11 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 20 | 11 | 31
  Between 18 and 65 years | 20 | 11 | 0 | 0 | 31
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.25 (4.82) | 32.64 (5.98) | 4.98 (.89) | 4.42 (.89) | 19.87 (15.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 9 | 4 | 43
  Male | 1 | 0 | 11 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 20 | 10 | 20 | 10 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 17 | 11 | 17 | 11 | 56
  More than one race | 2 | 0 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Child Glycemic Control
Description: Measure of hemoglobin A1c (HbA1c).
Time Frame: absolute value Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin cells
Groups:
- Standard of Care Control: Standard of Care: Parents in the standard of care control group will be instructed to manage their child's T1D as recommended by their diabetes team.
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
percentage of glycated hemoglobin cells | 7.56 (1.17) | 8.14 (0.73)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; repeated measures ANOVA; partial eta squared = .02

2. Primary Outcome: Parent Depressive Symptoms
Description: Center for Epidemiological Studies-Depression Scale Revised (CES-D); higher scores suggest worse outcome. Range 0-60.
Time Frame: absolute value Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
units on a scale | 10.0 (9.35) | 7.33 (8.28)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; repeated measures ANOVA; CESD-R = within subject variable; group = between subject variable; partial eta squared = .12

3. Primary Outcome: Parent Diabetes Distress
Description: Problem Areas in Diabetes Distress- Parent Report Questionnaire. Higher scores reflect worse outcome. Range 0-72
Time Frame: Absolute value at Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
units on a scale | 29.23 (18.86) | 27.36 (10.29)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; repeated measures ANOVA; partial eta squared = .03

4. Secondary Outcome: Family Mealtime behaviors_Frequency
Description: Behavioral Pediatrics Feeding Assessment Scale. This is a 35 item scale. This subscale reflects the frequency of perceived mealtime behavior problems (possible range: 35-175). Higher scores represent a worse outcome.
Time Frame: absolute value at Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
units on a scale | 78.23 (13.81) | 92.67 (14.93)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; repeated measures ANOVA; partial eta squared = .06

5. Secondary Outcome: Parents' Hypoglycemia Fear
Description: Measured using the Hypoglycemia Fear Survey (HFS-PYC). This is a 26 item measure and higher values represent a worse outcome. Range: 26-130.
Time Frame: absolute value at Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
units on a scale | 71.08 (15.96) | 64.00 (12.75)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; repeated measures ANOVA; partial eta squared = .04

6. Secondary Outcome: Parenting Stress- Frequency
Description: Measured using the Pediatric Inventory for Parents. This is a 42 item measure. Measure is scored so that higher values represent a worse outcome. Range: 42-210
Time Frame: Absolute value at Post-treatment (Week 33)
Population: lost to follow-up n=5 families in DIPPer group and n=2 families in standard care at 33 weeks; families withdrew themselves.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DIPPer Academy: Families randomized to this group will participate in the DIPPer Academy curriculum.
  DIPPer Academy: The DIPPer Academy curricula will build on treatment models guided by the Health Beliefs Model (HBM) and Social Cognitive Theory (SCT). The curricula includes video microlectures, personalize progress reports, and other features delivered via the internet.
- Standard of Care Control: DIPPer Academy: The DIPPer Academy curricula will build on treatment models guided by the Health Beliefs Model (HBM) and Social Cognitive Theory (SCT). The curricula includes video microlectures, personalize progress reports, and other features delivered via the internet.
  Standard of Care: Families in the standard of care control group will be instructed to manage their child's T1D as recommended.
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
units on a scale | 95.77 (32.78) | 90.44 (27.55)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; p < 0.05, repeated measures ANOVA; partial eta squared = .04

7. Secondary Outcome: Parents' T1D Self-efficacy
Description: Measured using the Parental Self-Efficacy Scale for Diabetes Management. This is an 8 item measure of self-efficacy. It has only a total score (items are summed for the total). Range 8-40. Higher scores represent a better outcome.
Time Frame: Absolute value at Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
units on a scale | 34.62 (3.91) | 33.67 (3.54)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; repeated measures ANOVA; partial eta squared = .24

8. Secondary Outcome: Parent Knowledge of T1D
Description: Test of Diabetes Knowledge-5. This is a 41 item measure. There is general knowledge (0-29) and Problem solving (0-11). This is scored based on percent of items correct, so higher scores represent a better outcome.
Time Frame: Absolute value at Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves.
Measure: Mean (Standard Deviation); unit: percentage of correct items
Arm/Group | DIPPer Academy | Standard of Care Control
Number analyzed (Participants) | 15 | 9
percentage of correct items | 98.94 (2.17) | 97.70 (2.99)
Statistical Analysis 1: Comparison: DIPPer Academy vs Standard of Care Control; Test type: Superiority; repeated measures ANOVA; partial eta squared = .03

9. Secondary Outcome: Behavioral Pediatric Feeding Assessment Scale_Problem
Description: Measured using the Behavioral Pediatrics Feeding Assessment Scale. This is a 35 item scale. This subscale reflects the number of mealtime behaviors that parents identify as problematic (possible range: 0-35). Higher scores represent a worse outcome.
Time Frame: Absolute value at Post-treatment (Week 33)
Population: lost to follow-up n=5 parents in DIPPer group and n=2 parents in standard care at 33 weeks; parents withdrew themselves.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DIPPer: Parents participating in DIPPer Academy
- Control: Parents receiving standard care
Arm/Group | DIPPer | Control
Number analyzed (Participants) | 15 | 9
score on a scale | 2.15 (2.85) | 7.18 (9.48)
Statistical Analysis 1: Comparison: DIPPer vs Control; Test type: Superiority; repeated measures ANOVA; partial eta squared = 0.04

ADVERSE EVENTS:
Time Frame: through study completion, average 7 months
Description: Definition for Serious Adverse Events and Adverse Events did not differ from clinicaltrials.gov definitions.
Groups:
- DIPPer Academy- Children: Parents randomized to this group will participate in the DIPPer Academy curriculum via the internet. Children did not receive treatment. We collected child HbA1c.
- Standard of Care Control- Children: Standard of Care: Parents in the standard of care control group will be instructed to manage their child's T1D as recommended by their diabetes team. We collected child HbA1c
Arm/Group | DIPPer Academy- Parents | Standard of Care Control- Parents | DIPPer Academy- Children | Standard of Care Control- Children
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/9 | 0/15 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/9 | 0/15 | 0/9
Other Adverse Events (participants affected / at risk) | 0/15 | 0/9 | 0/15 | 0/9

LIMITATIONS AND CAVEATS:
Small sample size leading to limited power to examine for treatment effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT03385265/Prot_SAP_001.pdf